CLINICAL TRIAL: NCT06558682
Title: Disitamab Vedotin Combined With Cisplatin for Neoadjuvant Therapy in Locally Advanced Cervical Cancer: a Prospective, Single-arm Clinical Trial
Brief Title: Neoadjuvant Therapy in Cervical Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: RemeGen Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kun Song, Chief Physician, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202405-012-1
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — disitamab vedotin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Disitamab Vedotin Combined with Cisplatin (Experimental): Locally advanced cervical cancer patient was treated with Disitamab Vedotin combined with Cisplatin for neoadjuvant therapy.
  Interventions: Drug: Disitamab Vedotin and Cisplatin

INTERVENTIONS:
Drug: Disitamab Vedotin and Cisplatin — Disitamab Vedotin: 2mg/Kg,ivdrip, 3 weeks/cycle,3 cycles. Cisplatin: 75-80mg/m2, ivdrip, 3 weeks/cycle,3 cycles.
  Other Names: Aidixi

SUMMARY:
In the comprehensive dataset of clinical diagnoses and treatments for cervical cancer in China, 49.8% of patients with stage IB3 and IIA2 receive surgical intervention following neoadjuvant chemotherapy. This indicates a pressing need to optimize neoadjuvant chemotherapy regimens for locally advanced cervical cancer. While paclitaxel combined with cisplatin is the conventional approach, 9.8% to 30.6% of patients demonstrate suboptimal responses, with a pathological complete response rate of approximately 10%.

Currently, the efficacy of antibody-drug conjugates in neoadjuvant chemotherapy for cervical cancer remains unexplored. This study seeks to address this gap by evaluating the combination of Disitamab Vedotin and Cisplatin in patients with stage IB3 and IIA2 cervical cancer with positive HER2 expression.The study will assess the impact of this regimen on pathological complete response rates, surgical complications, surgical resection rates, and overall survival.

DETAILED DESCRIPTION:
Primary research objectives:

To evaluate the effect of Disitamab Vedotin combined with cisplatin on pathological response rate (pCR) of locally advanced cervical cancer.

Secondary research objectives:

1. To evaluate the safety of Disitamab Vedotin combined with cisplatin;
2. To evaluate the effects of Disitamab Vedotin combined with cisplatin on surgical complications, surgical clearance rate and postoperative adjuvant treatment ratio;
3. To evaluate the effects of Disitamab Vedotin combined with cisplatin on objective tumor response rate (ORR), disease control rate (DCR) and survival;

Exploratory research objectives:

To explore the changes of tumor tissue protein expression, immune factors and HER-2 receptor expression before and after the use of ADC drugs, as well as biomarkers that can effectively predict the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cervical squamous cell carcinoma
* HER-2 positive

Exclusion Criteria:

* Cervical adenocarcinoma

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete remission | At the end of Cycle 3 (each cycle is 21 days)
  The rate of patients with pathological examination revealed an absence of malignant cells.

SECONDARY OUTCOMES:
Objective Response Rate | At the end of Cycle 3 (each cycle is 21 days)
  the proportion of patients whose tumor volume has shrunk to a predetermined value and maintains the minimum time frame required

CONTACTS AND LOCATIONS:
Overall Officials: Kun Song, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coleman RL, Lorusso D, Gennigens C, Gonzalez-Martin A, Randall L, Cibula D, Lund B, Woelber L, Pignata S, Forget F, Redondo A, Vindelov SD, Chen M, Harris JR, Smith M, Nicacio LV, Teng MSL, Laenen A, Rangwala R, Manso L, Mirza M, Monk BJ, Vergote I; innovaTV 204/GOG-3023/ENGOT-cx6 Collaborators. Efficacy and safety of tisotumab vedotin in previously treated recurrent or metastatic cervical cancer (innovaTV 204/GOG-3023/ENGOT-cx6): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2021 May;22(5):609-619. doi: 10.1016/S1470-2045(21)00056-5. Epub 2021 Apr 9. PMID 33845034
- [Background] Yonemori K, Kuboki Y, Hasegawa K, Iwata T, Kato H, Takehara K, Hirashima Y, Kato H, Passey C, Buchbjerg JK, Harris JR, Andreassen CM, Nicacio L, Soumaoro I, Fujiwara K. Tisotumab vedotin in Japanese patients with recurrent/metastatic cervical cancer: Results from the innovaTV 206 study. Cancer Sci. 2022 Aug;113(8):2788-2797. doi: 10.1111/cas.15443. Epub 2022 Jun 15. PMID 35633184
- [Background] Martinho O, Silva-Oliveira R, Cury FP, Barbosa AM, Granja S, Evangelista AF, Marques F, Miranda-Goncalves V, Cardoso-Carneiro D, de Paula FE, Zanon M, Scapulatempo-Neto C, Moreira MA, Baltazar F, Longatto-Filho A, Reis RM. HER Family Receptors are Important Theranostic Biomarkers for Cervical Cancer: Blocking Glucose Metabolism Enhances the Therapeutic Effect of HER Inhibitors. Theranostics. 2017 Jan 15;7(3):717-732. doi: 10.7150/thno.17154. eCollection 2017. PMID 28255362